CLINICAL TRIAL: NCT07034560
Title: Effectiveness of Oral Melatonin vs Oral Tranexamic Acid in the Treatment and Recurrence of Melasma : A Comparative, Randomized, Controlled Study
Brief Title: Effectiveness of Oral Melatonin vs Oral Tranexamic Acid in the Treatment and Recurrence of Melasma
Acronym: TXA-MELA
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Thammasat University (Other)
Responsible Party: Principal Investigator, Premjit Juntongjin, MD, Associate Professor, Principal Investigator, Thammasat University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CICM-MELASMA-MELATONIN-2025; MTU-EC-OO-0-238/67 (Other: Human Research Ethics Committee, Faculty of Medicine, Thammasat University)
Record Dates: First submitted 2025-06-10; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Melasma; Treatment Outcome; Recurrence
Keywords: Melasma; Hyperpigmentation; Tranexamic Acid; Melatonin; mMASI; Recurrence; Randomized Controlled Trial; Skin Pigmentation
MeSH Terms: conditions — Melanosis; Recurrence; Hyperpigmentation; Pigmentation Disorders | interventions — Tranexamic Acid; Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tranexamic Acid (TXA) (Active Comparator): Participants will receive 500 mg of oral tranexamic acid (Transamin®) once daily at bedtime for 12 weeks, along with a broad-spectrum sunscreen and a base cream.
  Interventions: Drug: Tranexamic Acid (TXA)
- melatonin (Circadin) (Experimental): Participants will receive 2 mg of oral melatonin (Circadin®) once daily at bedtime for 12 weeks, along with a broad-spectrum sunscreen and a base cream.
  Interventions: Drug: melatonin (Circadin)
- Placebo (Placebo Comparator): Participants will receive a placebo capsule once daily at bedtime for 12 weeks, along with a broad-spectrum sunscreen and a base cream.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tranexamic Acid (TXA) — 500 mg oral tranexamic acid (Transamin®), taken once daily at bedtime for 12 weeks.
  Arms: Tranexamic Acid (TXA)
Drug: melatonin (Circadin) — 2 mg oral melatonin (Circadin®), taken once daily at bedtime for 12 weeks.
  Arms: melatonin (Circadin)
Drug: Placebo — Placebo capsule identical in appearance, taken once daily at bedtime for 12 weeks.
  Arms: Placebo

SUMMARY:
This study compares the effectiveness of two oral medications-melatonin and tranexamic acid -in treating melasma, a common skin condition that causes dark facial patches.

Participants will be randomly assigned to receive either melatonin, tranexamic acid, or a placebo once daily at bedtime for 12 weeks. During this treatment phase, all participants will also apply a broad-spectrum sunscreen and a base cream.

After 12 weeks, participants will stop the oral medication but continue using the sunscreen and base cream for an additional 12 weeks to assess recurrence of melasma.

The study evaluates improvement in skin pigmentation, recurrence after treatment cessation, quality of life, and patient satisfaction.

This clinical trial will be conducted at Benchakitti Park Hospital, Bangkok, Thailand, and will enroll 75 adult participants.

DETAILED DESCRIPTION:
Melasma is a chronic skin disorder characterized by symmetrical, hyperpigmented patches on sun-exposed areas, especially the face. Although its exact cause is not fully understood, hormonal influences, ultraviolet (UV) exposure, and genetic predisposition are contributing factors.

Tranexamic acid (TXA), an antifibrinolytic agent, has shown promising results in treating melasma by inhibiting melanogenesis through the plasminogen-plasmin pathway. Melatonin (MLT), a hormone with antioxidant and anti-inflammatory properties, has also demonstrated potential benefits in melasma management by reducing oxidative stress and interfering with the melanin synthesis pathway.

This prospective, randomized, controlled, evaluator-blinded clinical trial aims to compare the efficacy and recurrence outcomes of oral TXA (500 mg), oral MLT (2 mg), and placebo, each administered once daily for 12 weeks. After discontinuing the oral treatment, all participants will continue using sunscreen and base cream for an additional 12 weeks to evaluate recurrence.

Outcome measures include modified Melasma Area and Severity Index (mMASI), Mexameter-based pigmentation indices, quality of life scores (DLQI), and patient satisfaction (VAS). The study is conducted at Benchakitti Park Hospital and includes 75 adult participants with epidermal or mixed-type melasma.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with the age above 18 years and above
2. Patients diagnosed with epidermal or mixed-type melasma

Exclusion Criteria:

1. Use of topical medications such as hydroquinone, whitening agents (e.g., arbutin, kojic acid, vitamin C, retinoids, and steroids) on melasma areas within 4 weeks prior to joining the study
2. Chemical peeling within 4 weeks prior to joining the study
3. Use of oral tranexamic acid or any supplements within 3 months prior to joining the study
4. History of laser treatment, dermabrasion, or skin-tightening devices within 6 months prior to joining the study
5. History of botulinum toxin injections, fillers, collagen stimulators, or thread lifts within 12 months prior to joining the study
6. Pregnancy or breastfeeding
7. Use of hormonal contraceptives within 1 year prior to joining the study
8. Personal or family history of thrombotic disorders, such as deep vein thrombosis, pulmonary embolism, stroke, protein C or S deficiency, or antithrombin III deficiency
9. History of more than 2 spontaneous abortion
10. History of impaired kidney function
11. History of cancer
12. Smoking
13. Heart disease (e.g., end-stage heart failure, chronic obstructive pulmonary disease, or use of prosthetic heart valves)
14. History of allergy to oral tranexamic acid or melatonin
15. Patients who are unable to follow up as per the study protocol
16. Patients with Hori's nevus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2024-11-12 (Actual); Primary Completion 2025-11-06 (Estimated); Study Completion 2025-11-06 (Estimated)

PRIMARY OUTCOMES:
Change in modified Melasma Area and Severity Index (mMASI) | Baseline, Week 4, Week 8, Week 12
  Change in modified Melasma Area and Severity Index (mMASI) score from baseline to Week 12.
  The mMASI ranges from 0 to 14.4, with higher scores indicating more severe melasma.
Change in modified Melasma Area and Severity Index (mMASI) (Recurrence) | Week 12, Week 16, Week 20, Week 24
  Recurrence is defined as an increase in mMASI score ≥50% from Week 12 to Week 24.
  The mMASI ranges from 0 to 14.4; higher scores indicate worse melasma.

SECONDARY OUTCOMES:
Melanin and Erythema Index | Baseline, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24
  Change in Melanin Index and Erythema Index at baseline to 24 weeks, measured by Mexameter.
  Higher values indicate increased pigmentation and erythema, respectively
Change in skin texture, pore size, fine line (Antera 3D imaging) | Baseline, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24
  Quantitative skin analysis using Antera 3D® imaging at baseline to 24 weeks. Lower scores indicate smoother texture, smaller pores, and fewer fine lines.
Dermatology Life Quality Index (DLQI) score | Baseline, Week 12, Week 24
  Change in Dermatology Life Quality Index (DLQI) from baseline to 24 weeks. DLQI ranges from 0 to 30. Higher scores indicate greater impairment in quality of life.
Patient satisfaction (Visual Analog Scale) | Baseline, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24
  Patient satisfaction score at every 4 weeks using Visual Analog Scale (VAS) from 0 to 10.
  Higher scores indicate greater satisfaction.
Adverse events (AEs) | Week 4, Week 8, Week 12
  Number and severity of treatment-emergent adverse events during the 12-week intervention

CONTACTS AND LOCATIONS:
Overall Officials: Assoc. Prof. Premjit Juntongjin, MD, Principal Investigator — Chulabhorn International College of Medicine, Thammasat University
Locations (1):
- Benchakitti Park Hospital, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to confidentiality concerns and lack of a formal data-sharing infrastructure. Data will be available upon reasonable request in de-identified, summary form only